CLINICAL TRIAL: NCT03574987
Title: The Effect of Dietary Carbohydrate Manipulation on All Major Aspects of Energy Balance: A 12-week Randomised Controlled Trial
Brief Title: Dietary Carbohydrate Manipulation and Energy Balance: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Dr, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHEB-Intervention
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Results first posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-01

CONDITIONS: Physical Activity; Diet Modification
Keywords: Physical Activity; Nutrition; Carbohydrates; Sugar; Energy Balance
MeSH Terms: conditions — Motor Activity | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with 3 arms. One arm is a typical diet (50% CHO, 20% SUG), one arm is low sugar (50% CHO, <5% SUG), one arm is low carbohydrate (<8% CHO, <5% SUG). Stratified by sex and physical activity level (PAL).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL (Active Comparator): Diet consisting of 50% carbohydrate (20% sugar), 15% protein, 35% fat
  Interventions: Other: Diet
- LOW SUG (Experimental): Diet consisting of 50% carbohydrate (<5% sugar), 15% protein, 35% fat
  Interventions: Other: Diet
- LOW CHO (Experimental): Diet consisting of <8% carbohydrate (<5% sugar), 15% protein, >77% fat
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Macronutrient composition (specifically type and/or amount of carbohydrate) is manipulated

SUMMARY:
This study will investigate how dietary sugar and carbohydrates influence metabolism and health across a 12-week period, with a focus on physical activity. One third of participants will eat a diet with typical amounts of sugar and carbohydrate, one third of participants will eat a diet with sugar intake restricted, and the final third of participants will eat a diet where both sugar and total carbohydrates are restricted and replaced with fat.

DETAILED DESCRIPTION:
Sugar is perceived negatively, leading to government taxation and targets to reduce consumption. These actions have been taken based on the limited evidence that high-sugar diets are associated with greater total energy intake. However, energy intake is only one half of the energy balance equation (energy in vs energy out). Without considering energy expenditure, it is impossible to fully understand the effects of sugar on health. Removing dietary sugar or carbohydrates from the diet may influence energy balance through mechanisms other than energy intake - for example by reducing levels of physical activity.

Understanding dietary regulators of energy balance is more important than ever because diseases like obesity are a consequence of energy surplus (i.e. energy in > energy out). No studies have investigated a causal role of dietary sugar or carbohydrate on energy balance. The proposed research will seek to understand the responses to manipulating dietary carbohydrate and sugar content on energy balance and health. This research will enable the public to make informed dietary choices about carbohydrate and sugar consumption.

To achieve this, healthy non-obese adults, aged 18-65 years will be recruited to take part in an intervention study with measures of energy intake, energy expenditure, metabolic health, gut microbiota, and appetite. All laboratory trials will take place at the University of Bath. Participants will be randomised to consume one of three diets for a period of 12 weeks, with laboratory visits at baseline, at week 4, and at week 12:

1. CONTROL (moderate sugar) - reflecting the composition of a typical European diet
2. Low sugar - the same composition of a typical European diet but with <5% energy intake from sugar
3. Low carbohydrate - low carbohydrate diet with <5% energy intake from sugar, replacing carbohydrate energy with fat

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5-29.9 kg∙m-2
* Age 18-65 years
* Able and willing to provide informed consent and safely comply with study procedures
* Females to maintain record of regular menstrual cycle phase/contraceptive use
* No anticipated changes in physical activity during the first 4 weeks of the study (e.g. holidays or training programmes)

Exclusion Criteria:

* Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias
* Any diagnosed metabolic disease (e.g. type 1 or type 2 diabetes)
* Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment
* Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)
* Any reported recent (<6 months) change in body mass (± 3%)
* Use of antibiotic medication in the last 3 months
* Use of prebiotic or probiotic products in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith HA, Gonzalez JT, Thompson D, Betts JA. Dietary carbohydrates, components of energy balance, and associated health outcomes. Nutr Rev. 2017 Oct 1;75(10):783-797. doi: 10.1093/nutrit/nux045. PMID 29028272
- [Background] Betts JA, Richardson JD, Chowdhury EA, Holman GD, Tsintzas K, Thompson D. The causal role of breakfast in energy balance and health: a randomized controlled trial in lean adults. Am J Clin Nutr. 2014 Aug;100(2):539-47. doi: 10.3945/ajcn.114.083402. Epub 2014 Jun 4. PMID 24898233
- [Background] Erickson J, Sadeghirad B, Lytvyn L, Slavin J, Johnston BC. The Scientific Basis of Guideline Recommendations on Sugar Intake: A Systematic Review. Ann Intern Med. 2017 Feb 21;166(4):257-267. doi: 10.7326/M16-2020. Epub 2016 Dec 20. PMID 27992898
- [Derived] Bergwall S, Johansson A, Sonestedt E, Acosta S. High versus low-added sugar consumption for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2022 Jan 5;1(1):CD013320. doi: 10.1002/14651858.CD013320.pub2. PMID 34986271

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CONTROL | LOW SUG | LOW CHO
Started | 20 | 18 | 22
Completed | 13 | 16 | 16
Not Completed | 7 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CONTROL | LOW SUG | LOW CHO | Total
Number analyzed (Participants) | 18 | 17 | 18 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (18) | 32 (16) | 34 (14) | 35 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 9 | 30
  Male | 7 | 7 | 9 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18 | 17 | 18 | 53

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Energy Expenditure (kJ/Day or kcal/Day)
Description: 24-hour physical activity energy expenditure (kJ/day or kcal/day)
Time Frame: 7 days (across 12 weeks) - Primary outcome at week 4
Population: Dropout and/or missing data (device malfunction) between weeks 4 and 12.
Measure: Mean (95% Confidence Interval); unit: kcal/d
Arm/Group | CONTROL | LOW SUG | LOW CHO
Number analyzed (Participants) | 17 | 16 | 16
kcal/d
  Week 4 | 1229 [1066 to 1392] | 1096 [929 to 1263] | 1275 [1107 to 1442]
  Week 12: number analyzed (Participants) | 12 | 15 | 13
  Week 12 | 1142 [959 to 1324] | 1077 [914 to 1240] | 1136 [960 to 1311]

2. Secondary Outcome: Time Spent in Different Physical Activity Intensities (MET Categories) (Minutes)
Description: Time spent in different physical activity intensities (MET categories) (minutes)
Time Frame: 7 days (across 12 weeks)
Reporting Status: Not Posted

3. Secondary Outcome: Energy Expended in Different Physical Activity Intensities (MET Categories) (kJ or kcal)
Description: Energy expended in different physical activity intensities (MET categories) (kJ or kcal)
Time Frame: 7 days (across 12 weeks)
Reporting Status: Not Posted

4. Secondary Outcome: Energy Intake and Dietary Macronutrient Composition
Description: Estimated using food diaries, 7 days each time concurrently measured with PAEE and 3 days per week for the rest of the intervention
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Body Mass
Description: Measured weekly using electric scales
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Bone Mineral Density
Description: Bone mineral density measured using dual x-ray absorptiometry
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Bone Mineral Content
Description: Bone mineral content measured using dual x-ray absorptiometry
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Fat Mass
Description: Fat mass measured using dual x-ray absorptiometry
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Fat-free Mass
Description: Fat-free mass measured using dual x-ray absorptiometry
Time Frame: 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Android Fat Mass
Description: Android fat mass measured using dual x-ray absorptiometry
Time Frame: 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Gynoid Fat Mass
Description: Gynoid fat mass measured using dual x-ray absorptiometry
Time Frame: 12 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Resting Metabolic Rate
Description: Resting metabolic rate will be measured using indirect calorimetry
Time Frame: 12 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Substrate Oxidation
Description: Substrate oxidation will be measured using indirect calorimetry both at rest and during exercise
Time Frame: 12 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Waist and Hip Circumference
Description: Waist and hip circumference will be measured using a tape measure
Time Frame: 12 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Step Count
Description: Measured daily using pedometers
Time Frame: 12 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Fasting Metabolite/Hormone Profile
Description: Assessment of blood glucose, insulin, triglycerides, non-esterified fatty acids, lactate, beta-hydroxybutyrate, leptin, fibroblast growth factor-21, total cholesterol, high density lipoprotein, and low density lipoprotein concentrations, appetite hormone concentrations (including PYY, GLP-1, ghrelin)
Time Frame: 12 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Postprandial Metabolite/Hormone Profile
Description: as for outcome 16
Time Frame: 4 hours (across 12 weeks)
Reporting Status: Not Posted

18. Secondary Outcome: Blood Pressure
Description: Measured using an automated sphygmomanometer
Time Frame: 12 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Food Preference Ratings
Description: Food preference ratings determined by bespoke computer software
Time Frame: 12 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Subjective Appetite and Mood Ratings
Description: Measured by 0-100 mm visual analogue scale
Time Frame: 12 weeks
Reporting Status: Not Posted

21. Secondary Outcome: Interstitial Glucose Concentrations
Description: Measured using research-grade freestyle libre glucose monitors. Measured pre-, during- and at the end of the intervention
Time Frame: 14 days (across 12 weeks)
Reporting Status: Not Posted

22. Secondary Outcome: Adipose Tissue Gene Expression
Description: Expression of a panel of genes related to glucose metabolism in adipose biopsies using real-time polymerase chain reaction
Time Frame: 12 weeks
Reporting Status: Not Posted

23. Secondary Outcome: Adipose Tissue Protein Expression
Description: Expression of various proteins related to glucose metabolism in adipose biopsies via Western blot
Time Frame: 12 weeks
Reporting Status: Not Posted

24. Secondary Outcome: Muscle Tissue Gene Expression
Description: Expression of a panel of genes related to glucose metabolism in muscle biopsies using real-time polymerase chain reaction
Time Frame: 12 weeks
Reporting Status: Not Posted

25. Secondary Outcome: Muscle Tissue Protein Expression
Description: Expression of various proteins related to glucose metabolism in muscle biopsies via Western blot
Time Frame: 12 weeks
Reporting Status: Not Posted

26. Secondary Outcome: Muscle Glycogen Concentrations
Description: Glycogen concentrations measured from vastus lateralis muscle samples
Time Frame: 12 weeks
Reporting Status: Not Posted

27. Secondary Outcome: Gut Microbiome Characterisation
Description: Faecal sample DNA and water will be used to determine taxonomic and functional diversity of microbes using transcriptomic techniques
Time Frame: 12 weeks
Reporting Status: Not Posted

28. Secondary Outcome: Urinary Acetoacetate Concentrations
Description: Will be measured using handheld sticks
Time Frame: 12 weeks
Reporting Status: Not Posted

29. Secondary Outcome: Urine Urea Nitrogen Excretion
Description: Will be measured across trial days
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | CONTROL | LOW SUG | LOW CHO
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CONTROL (N=18) | LOW SUG (N=17) | LOW CHO (N=18)
Sports injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03574987/Prot_SAP_000.pdf